CLINICAL TRIAL: NCT05034809
Title: Effectiveness Of High Dose Melatonin As Adjunctive Therapy For Pediatric Patients Diagnosed With Dengue Fever With Warning Signs: A Randomized Control Trial
Brief Title: Effectiveness Of High Dose Melatonin As Adjunctive Therapy For Dengue Fever With Warning Signs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ilocos Training and Regional Medical Center (Other Government)
Responsible Party: Principal Investigator, Navid Roodaki, Pediatric Chief Resident, Ilocos Training and Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITRMC-REC-2020-045
Record Dates: First submitted 2021-08-22; First posted 2021-09-05 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Dengue Fever With Warning Signs
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator
Masking Description: The research assistant will explain to the parents and to the child if capable of understanding the clinical trial. However, the participants, family and the researcher will not know until the end of the study if they were placed in the control group or treatment group. Blinding will be done using a pre-generated number code and QR code which, when scanned by the research assistant at the end of the study, it will reveal to what group the patient was randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Other than the guided management of Dengue Fever with warning signs, the treatment group will receive a standard dose of 20mg/day of melatonin20-21 for 5 days. The dosing was based on the study by Leiberman et al and Malhotra et al. If a patient is unable to tolerate the whole or punctured tablet, it will be given with milk or water. There is no known interaction between melatonin and milk known to date. Daily complete blood count will be done and be recording in an electronic record using Microsoft Excel.
  Interventions: Drug: Melatonin 20 MG
- Control Group (No Intervention): Other than the guided management of Dengue Fever with warning signs, the control group will be manage according the Department of Health Dengue Management Guideline. No placebo will be given.

INTERVENTIONS:
Drug: Melatonin 20 MG — Melatonin, also known as N-acetyl-5-methoxytryptamine will be the main intervention given to participating patients of this study. This study will use a dose of 20mg/day using the commercially available 5mg/tablet20-21. If a patient cannot be tolerate swallowing the whole tablet, it will be crushed and mixed with milk. According to the study done by Shah et al. there was no degradation in the active component of melatonin when mixed with milk or food as a medium for drug delivery.
  Arms: Treatment Group

SUMMARY:
Dengue Hemorrhagic Fever is a mosquito-borne viral disease endemic in the Philippines which caused multiple epidemics. Most points to the activation of the complement system secondary to humoral respond leading to cytokine release causing systemic inflammation. Melatonin, is a hormone which has an a) anti-viral, b) immunomodulator, c) antioxidant, d) modulatory effect on hematopoiesis and e) anti-inflammatory action.

This is a randomized control trial to determine the effectiveness of adjunctive melatonin therapy among patients diagnosed with Dengue fever with Warning Signs. This would include children aged 5 to 18 years old with no signs of hemmorhagic shock. They would be randomly assigned into 2 groups. Baseline Complete blood count with platelet (CBCPC) will be collected. Daily CBCPC will be collected and would be statistically analyze after the study.

DETAILED DESCRIPTION:
Dengue Hemorrhagic Fever is a mosquito-borne viral disease endemic in the Philippines which caused multiple epidemics. Most points to the activation of the complement system secondary to humoral respond leading to cytokine release causing systemic inflammation. Melatonin, is a hormone which has an a) anti-viral, b) immunomodulator, c) antioxidant, d) modulatory effect on hematopoiesis and e) anti-inflammatory action.

Main Objective:

To determine the effectiveness of Melatonin tablet as an adjunctive therapy in decreasing morbidity for pediatric patients diagnosed with Dengue Fever with Warning Signs at Ilocos Training and Regional Medical Center Department of Pediatrics.

Specific Objective

1. To determine the clinical profiles of pediatric patients diagnosed with Dengue Fever with Warning Signs in Ilocos Training and Regional Medical Center
2. To determine the effectiveness of Melatonin 20mg as adjunctive therapy for pediatric patients diagnosed with Dengue Fever with Warning Signs with regards to:

   a. Number of days for resolution of fever from the 1st day of administration of melatonin b. Number of days for the platelet count to increase from the 1st day of administration of melatonin c. Number of days for the white blood cell count to increase from the 1st day of administration of melatonin d. Absence of subsequent complications in the critical phase of the illness (4th - 6th day of illness) i. Presence of mucosal bleeding, melena, epistaxis ii. Presence of ascites, pleural effusion, edema iii. Hypotension, tachycardia iv. Increase capillary refill time

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient aged 5 to 18 years old with febrile episodes (Temperature >/= 37.8 degrees Celsius) with positive Dengue NS1.

  2. Patients with Dengue Fever on the Department of Health 2012 definition of Dengue fever with Warning Signs with any one of the following:
  1. Abdominal tenderness
  2. Persistent vomiting
  3. Minimal mucosal bleed
  4. Platelet count less than or equal to 100,000

     Exclusion Criteria:
* 1. Patients with signs and symptoms related to dengue fever but with negative Dengue Ns1 result.

  2. Patients diagnosed as Severe Dengue or Dengue Shock. 3. Patients unable to tolerate tablet formulation. 4. Patients placed on nothing per Orem. 5. Patients previously treated in a referring facility.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Number Of Days Prior To Elevation of Platelet Count Among Dengue Fever with Warningn Signs Patient Given Melatonin 20mg. | 1 year
  Effectiveness Of Melatonin Tablet As An Adjunctive Therapy In Decreasing Morbidity For Pediatric Patients Diagnosed With Dengue Fever With Warning Signs

SECONDARY OUTCOMES:
Incidence Of Dengue Fever with Warning Signs among Pediatric Population at Ilocos Training and Regional Medical Center. | 1 year
  Clinical Profiles Of Pediatric Patients Diagnosed With Dengue Fever With Warning Signs In Ilocos Training And Regional Medical Center
determine the effectiveness of Melatonin 20mg as adjunctive therapy for pediatric patients diagnosed with Dengue Fever with Warning Signs | 1 year
  1. Number of days for the platelet count to increase from the 1st day of administration of melatonin
  2. Number of days for the white blood cell count to increase from the 1st day of administration of melatonin
  3. Absence of subsequent complications in the critical phase of the illness (4th - 6th day of illness)
  i. Presence of mucosal bleeding, melena, epistaxis ii. Presence of ascites, pleural effusion, edema iii. Hypotension, tachycardia iv. Increase capillary refill time
Number Of Days Prior To Elevation of White Blood Cells Among Dengue Fever with Warningn Signs Patient Given Melatonin 20mg. | 1 year
  Effectiveness Of Melatonin Tablet As An Adjunctive Therapy In Decreasing Morbidity For Pediatric Patients Diagnosed With Dengue Fever With Warning Signs

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Lydia O Ramirez, MD, Study Chair — Ilocos Training and Regional Medical Center

IPD SHARING:
Plan to Share IPD: No
Due to the Data Privacy Act of the Philippines, only the completed data will be shared